Date: 07/22/2024

National Clinical Trials #: NCT04637815

Study Title: A Social Network AOD Intervention for Homeless Youth Transitioning to Housing

#### I. WHAT IS THIS STUDY ABOUT?

The Village Family Services (TVFS) is partnering with RAND, which is a non-profit research organization in Santa Monica, on a research project to evaluate a social network tool to assist new residents of housing programs who have used alcohol or drugs in the past year. This social network tool is designed to help new residents make healthy choices in terms of alcohol and drug use, as well as strengthen their supportive connections with others. We are asking you and about 60 other young adults to participate. The research project is paid for by the National Institute on Drug Abuse.

## II. WHAT WILL WE ASK YOU TO DO?

The services you receive at TVFS will be the same whether or not you help us test the new program. If you want to participate in the project, you will be asked to do two things:

- **1. Complete two phone surveys**. The surveys will ask you about your social networks, alcohol and drug use, and other recent behaviors. Each survey will take about 30-45 minutes to complete. The first survey will take place soon and the next one will be 3 months from now. Your answers are confidential. **We will pay you a \$30 for the first survey and \$40 for the second survey.**
- 2. Meet regularly with your case manager. RAND will randomly choose some people to use the social network tool with their case manager four times over the next two months, and some people to meet with their case manager as usual over the next two months. This means that you will have an equal chance of being part of the social network case management meetings or regular case management meetings. If you are selected to receive the social network case management, you will share and receive information about your social network. Regardless of which group you are in, you will receive a \$5 gift card for each of the four case management meetings you attend as part of this project.

## III. COSTS

• You do not have to pay money to be part of this project. The services you receive at TVFS will be the same whether or not you decide to be part of this project.

## **IV. BENEFITS**

 Your participation will help us improve case management services for new residents of housing programs.

## V. RISKS

 Some of the questions you will be asked on the survey or during case management may make you feel uncomfortable. You can choose not to answer questions and you may leave the session or stop the survey at any time.

## VI. CONFIDENTIALITY

To help us protect your privacy, we have obtained a Confidentiality Certificate from the Department of Health and Human Services (DHHS). This certificate says that RAND does not have to tell anyone any information about you. This includes any civil, criminal, administrative, legislative, or other proceedings, whether State, Federal, or local. The Certificate does not imply approval or disapproval of the project by the Secretary of DHHS. You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, medical care provider, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

<u>Your confidentiality is very important to us.</u> We will not write your name, address or any other information about you on your materials. We will give you an ID number to protect your confidentiality. We will only share your information with other RAND project staff helping with this study. We will not share your information with your employer, family members or law enforcement officials.

There are only two times where we might need to tell others about your information. We will only tell others about your information if:

- 1. We need to keep you and other people safe. An example of this is if you want to hurt yourself or others. In that case, we will give information about you to others (e.g., 911, research staff), including TVFS program staff, in order to keep you and other people safe.
- 2. You tell us about someone hurting a child or an elderly person. In that case, we must report it to TVFS staff, who may report it to the authorities.

The four sessions that you have with your case manager as part of this project will be audio recorded. This is for quality assurance purposes only; that is, we want to ensure that the sessions go as planned. No one outside of the RAND project staff helping with this study will be able to listen to these recorded sessions. We will destroy all audio recordings at the end of the project.

## VII. YOUR PARTICIPATION

You do not have to be part of this project and are free to withdraw from the project at any time. Your choice does not affect the services you receive at TVFS or anywhere else. You may leave the project at any time and you will still be able to meet with your case manager. You can skip any questions that you do not want to answer on the survey or during the case management meetings as part of this project.

## **VIII. WHO IS LEADING THE PROJECT?**

Dr. David Kennedy from RAND is leading the project. If you have any questions or want to talk to us, please call Dr. Kennedy at 1-800-447-2631, ext. 6133.

## IX. IF YOU HAVE QUESTIONS

If you have questions about your rights as a research participant, you can contact RAND's Human Subjects Protection Committee toll-free at (866) 697-5620 or by emailing <a href="mailto:hspcinfo@rand.org">hspcinfo@rand.org</a>. If possible, when you contact the Committee, please reference Study # 2018-0529.

| TO BE COMPLETED BY GRAY INSIGHT STAFF ONLY: | |
|---|---|
| I have read the information in this document to the individual named above. S/he has indicated that they understand the information and agree to participate in this project. | |
| Name (please print): | |
| Signature: | Date: |

To be completed by Gray Insight staff:

| PLEASE CONTACT ME ABOUT THIS RESEARCH PROJECT: | |
|---|---|
| 1. | Name (please print): |
| 2. | Best phone number to reach me: () |
| 3. | Another phone number where I can be reached: () |
| 4. | Best days to reach me: (CIRCLE ALL THAT APPLY) |
| | Monday Tuesday Wednesday Thursday Friday Saturday Sunday |
| 5. | Best times to reach me: Mornings Afternoons Evenings |
| 6. | Signature: Date: |